CLINICAL TRIAL: NCT00839241
Title: An Open , Prospective, Randomized, Parallel Group Study to Investigate Whether Postoperatively Collected and Transfused Autologous Whole Blood Improves the Immunological Status in Comparison to Allogenic Blood Transfusion in Patients Undergoing Total Knee Replacement
Brief Title: A Clinical Study to Investigate if Transfusion of Patients Own Shed Blood Improves the Immunological Status in Comparison to Transfusion of Donor Blood ("Bank Blood")
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wellspect HealthCare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YA-ABT-0004
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Results first posted 2010-10-04 (Estimated); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Arthroplasty, Replacement, Knee; Blood Transfusion, Autologous; Blood Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Autologous Blood Transfusion (Experimental)
  Interventions: Device: Bellovac ABT
- Allogenic Blood Transfusion (Active Comparator)
  Interventions: Procedure: Allogenic Blood Transfusion

INTERVENTIONS:
Device: Bellovac ABT — Bellovac ABT (autologous blood)
  Arms: Autologous Blood Transfusion
Procedure: Allogenic Blood Transfusion — Transfusion of allogenic ("bank") blood.
  Arms: Allogenic Blood Transfusion

SUMMARY:
The primary objective of the study is to compare the immunological status after either autologous blood transfusion as administered by Bellovac® ABT or allogenic blood transfusion, with regards to change in Natural Killer (NK) cell frequency in patients undergoing total knee replacement.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Male and female patients aged 18 years and over scheduled for total knee replacement
* Subjects classified as ASA Physical Status Classification System class P1, P2 or P3 according to the American Society of Anaesthesiology

Exclusion Criteria:

* Involvement in the planning and conduct of the study (applies to both Astra Tech staff or staff at the study site)
* Pre-operatively haemoglobin below normal range as judged by the investigator
* Previous enrolment or randomisation to treatment in the present study
* Expected or confirmed participation in another clinical study during the study period
* Severe non-compliance to protocol as judged by the investigator and/or Astra Tech
* Current symptoms of haemophilia
* History of or presence of malignant disease with propensity for systemic spread during the last 5 years
* Current or expected use of cytotoxic drugs
* Current untreated anaemia (e.g. sickle cell anaemia) as deemed by investigator
* Use of pre-donation
* Use of recombinant erythropoetin
* Use of other autologous blood transfusion than that with Bellovac ABT, e.g. washed and centrifuged blood like CellSaver

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Jacobsson, MD, PhD, Prof., Study Director — Dentsply Sirona Implants and Consumables
Locations (1):
- Specjalistyczny Szpital Im. Alfreda Sokolowskiego, Szczecin, Poland

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Autologous Blood Transfusion | Allogenic Blood Transfusion
Started | 20 | 25
Completed | 15 | 8
Not Completed | 5 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Autologous Blood Transfusion | Allogenic Blood Transfusion | Total
Number analyzed (Participants) | 20 | 25 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 12 | 19
  >=65 years | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (10.3) | 66.6 (8.3) | 66.8 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 20 | 33
  Male | 7 | 5 | 12
Region of Enrollment [Number; unit: participants]
  Poland | 20 | 25 | 45

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Natural Killer Cells as Measured With Flow Cytometry.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: total number of cells * 10^5/mL
Arm/Group | Autologous Blood Transfusion | Allogenic Blood Transfusion
Number analyzed (Participants) | 20 | 25
total number of cells * 10^5/mL | 2.98 (1.62) | 2.26 (1.13)

2. Primary Outcome: Frequency of Natural Killer Cells as Measured With Flow Cytometry.
Time Frame: Day 5 postop
Measure: Mean (Standard Deviation); unit: total number of cells * 10^5/mL
Arm/Group | Autologous Blood Transfusion | Allogenic Blood Transfusion
Number analyzed (Participants) | 20 | 25
total number of cells * 10^5/mL | 2.79 (2.11) | 1.96 (1.19)

3. Primary Outcome: Frequency of Natural Killer Cells as Measured With Flow Cytometry.
Time Frame: Day 8 postop
Measure: Mean (Standard Deviation); unit: total number of cells * 10^5/mL
Arm/Group | Autologous Blood Transfusion | Allogenic Blood Transfusion
Number analyzed (Participants) | 20 | 25
total number of cells * 10^5/mL | 2.80 (2.03) | 1.79 (0.94)

4. Primary Outcome: Natural Killer Cells (Proportion of Lymphocytes, Measured With Flow Cytometry)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Autologous Blood Transfusion | Allogenic Blood Transfusion
Number analyzed (Participants) | 20 | 25
Percent | 13.8 (6.3) | 12.3 (4.6)

5. Primary Outcome: Natural Killer Cells (Proportion of Lymphocytes, Measured With Flow Cytometry)
Time Frame: Day 5 postop
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Autologous Blood Transfusion | Allogenic Blood Transfusion
Number analyzed (Participants) | 20 | 25
Percent | 12.1 (5.3) | 9.3 (4.3)

6. Primary Outcome: Natural Killer Cells (Proportion of Lymphocytes, Measured With Flow Cytometry)
Time Frame: Day 8 postop
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Autologous Blood Transfusion | Allogenic Blood Transfusion
Number analyzed (Participants) | 20 | 25
Percent | 11.5 (5.6) | 7.4 (2.5)

7. Secondary Outcome: Interferon Gamma
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Autologous Blood Transfusion | Allogenic Blood Transfusion
Number analyzed (Participants) | 20 | 25
pg/mL | 5.6 (2.6) | 6.2 (4.2)

8. Secondary Outcome: Interferon Gamma
Time Frame: Day 5 postop
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Autologous Blood Transfusion | Allogenic Blood Transfusion
Number analyzed (Participants) | 20 | 25
pg/mL | 6.5 (2.1) | 5.5 (3.8)

9. Secondary Outcome: Interferon Gamma
Time Frame: Day 8 postop
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Autologous Blood Transfusion | Allogenic Blood Transfusion
Number analyzed (Participants) | 20 | 25
pg/mL | 6.25 (2.5) | 6.99 (4.8)

10. Secondary Outcome: Interleukin-2
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Autologous Blood Transfusion | Allogenic Blood Transfusion
Number analyzed (Participants) | 20 | 25
pg/mL | 6.3 (3.3) | 8.4 (6.9)

11. Secondary Outcome: Interleukin-2
Time Frame: Day 5 postop
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Autologous Blood Transfusion | Allogenic Blood Transfusion
Number analyzed (Participants) | 20 | 25
pg/mL | 6.4 (3.6) | 8.0 (6.7)

12. Secondary Outcome: Interleukin-2
Time Frame: Day 8 postop
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Autologous Blood Transfusion | Allogenic Blood Transfusion
Number analyzed (Participants) | 20 | 25
pg/mL | 7.1 (5.5) | 8.8 (7.1)

13. Secondary Outcome: Interleukin-4
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Autologous Blood Transfusion | Allogenic Blood Transfusion
Number analyzed (Participants) | 20 | 25
pg/mL | 4.9 (2.2) | 6.1 (4.7)

14. Secondary Outcome: Interleukin-4
Time Frame: Day 5 postop
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Autologous Blood Transfusion | Allogenic Blood Transfusion
Number analyzed (Participants) | 20 | 25
pg/mL | 5.5 (2.2) | 5.4 (4.4)

15. Secondary Outcome: Interleukin-4
Time Frame: Day 8 postop
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Autologous Blood Transfusion | Allogenic Blood Transfusion
Number analyzed (Participants) | 20 | 25
pg/mL | 5.5 (3.5) | 6.2 (4.4)

16. Secondary Outcome: Interleukin-6
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Autologous Blood Transfusion | Allogenic Blood Transfusion
Number analyzed (Participants) | 20 | 25
pg/mL | 6.1 (2.9) | 7.0 (4.9)

17. Secondary Outcome: Interleukin-6
Time Frame: Day 5 postop
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Autologous Blood Transfusion | Allogenic Blood Transfusion
Number analyzed (Participants) | 20 | 25
pg/mL | 10.5 (2.8) | 14.0 (7.8)

18. Secondary Outcome: Interleukin-6
Time Frame: Day 8 postop
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Autologous Blood Transfusion | Allogenic Blood Transfusion
Number analyzed (Participants) | 20 | 25
pg/mL | 9.1 (4.2) | 12.5 (3.6)

19. Secondary Outcome: Interleukin-10
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Autologous Blood Transfusion | Allogenic Blood Transfusion
Number analyzed (Participants) | 20 | 25
pg/mL | 5.8 (3.9) | 8.0 (6.2)

20. Secondary Outcome: Interleukin-10
Time Frame: Day 5 postop
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Autologous Blood Transfusion | Allogenic Blood Transfusion
Number analyzed (Participants) | 20 | 25
pg/mL | 7.5 (3.4) | 7.9 (5.7)

21. Secondary Outcome: Interleukin-10
Time Frame: Day 8 postop
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Autologous Blood Transfusion | Allogenic Blood Transfusion
Number analyzed (Participants) | 20 | 25
pg/mL | 6.5 (4.1) | 8.9 (6.2)

22. Secondary Outcome: TNF-Alpha
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Autologous Blood Transfusion | Allogenic Blood Transfusion
Number analyzed (Participants) | 20 | 25
pg/mL | 6.7 (2.9) | 8.0 (6.3)

23. Secondary Outcome: TNF-Alpha
Time Frame: Day 5 postop
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Autologous Blood Transfusion | Allogenic Blood Transfusion
Number analyzed (Participants) | 20 | 25
pg/mL | 7.1 (3.4) | 7.4 (5.4)

24. Secondary Outcome: TNF-Alpha
Time Frame: Day 8 postop
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Autologous Blood Transfusion | Allogenic Blood Transfusion
Number analyzed (Participants) | 20 | 25
pg/mL | 7.6 (3.4) | 8.0 (5.7)

25. Secondary Outcome: Hemoglobin
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Autologous Blood Transfusion | Allogenic Blood Transfusion
Number analyzed (Participants) | 20 | 25
g/dL | 14.5 (1.0) | 13.3 (1.3)

26. Secondary Outcome: Hemoglobin
Time Frame: Day 1 postop
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Autologous Blood Transfusion | Allogenic Blood Transfusion
Number analyzed (Participants) | 20 | 25
g/dL | 11.7 (0.9) | 11.0 (1.5)

27. Secondary Outcome: Hemoglobin
Time Frame: Day 5 postop
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Autologous Blood Transfusion | Allogenic Blood Transfusion
Number analyzed (Participants) | 20 | 25
g/dL | 11.1 (1.5) | 10.5 (1.5)

28. Secondary Outcome: Hemoglobin
Time Frame: Day 8 postop
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Autologous Blood Transfusion | Allogenic Blood Transfusion
Number analyzed (Participants) | 20 | 25
g/dL | 11.1 (1.4) | 10.6 (1.0)

29. Secondary Outcome: Erythrocyte Volume Fraction
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: percentage of blood volume
Arm/Group | Autologous Blood Transfusion | Allogenic Blood Transfusion
Number analyzed (Participants) | 20 | 25
percentage of blood volume | 45.1 (2.4) | 41.3 (3.3)

30. Secondary Outcome: Erythrocyte Volume Fraction
Time Frame: Day 1 postop
Measure: Mean (Standard Deviation); unit: percentage of blood volume
Arm/Group | Autologous Blood Transfusion | Allogenic Blood Transfusion
Number analyzed (Participants) | 20 | 25
percentage of blood volume | 36.1 (2.7) | 33.8 (4.3)

31. Secondary Outcome: Erythrocyte Volume Fraction
Time Frame: Day 5 postop
Measure: Mean (Standard Deviation); unit: percentage of blood volume
Arm/Group | Autologous Blood Transfusion | Allogenic Blood Transfusion
Number analyzed (Participants) | 20 | 25
percentage of blood volume | 34.7 (4.6) | 32.8 (4.9)

32. Secondary Outcome: Erythrocyte Volume Fraction
Time Frame: Day 8 postop
Measure: Mean (Standard Deviation); unit: percentage of blood volume
Arm/Group | Autologous Blood Transfusion | Allogenic Blood Transfusion
Number analyzed (Participants) | 20 | 25
percentage of blood volume | 35.1 (3.8) | 33.3 (3.4)

33. Secondary Outcome: Leucocyte Particle Concentration
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: 10^3/uL
Arm/Group | Autologous Blood Transfusion | Allogenic Blood Transfusion
Number analyzed (Participants) | 20 | 25
10^3/uL | 5.8 (1.3) | 5.3 (1.6)

34. Secondary Outcome: Leucocyte Particle Concentration
Time Frame: Day 1 postop
Measure: Mean (Standard Deviation); unit: 10^3/uL
Arm/Group | Autologous Blood Transfusion | Allogenic Blood Transfusion
Number analyzed (Participants) | 20 | 25
10^3/uL | 9.4 (3.0) | 7.3 (2.3)

35. Secondary Outcome: Leucocyte Particle Concentration
Time Frame: Day 5 postop
Measure: Mean (Standard Deviation); unit: 10^3/uL
Arm/Group | Autologous Blood Transfusion | Allogenic Blood Transfusion
Number analyzed (Participants) | 20 | 25
10^3/uL | 6.7 (1.8) | 6.1 (2.2)

36. Secondary Outcome: Leucocyte Particle Concentration
Time Frame: Day 8 postop
Measure: Mean (Standard Deviation); unit: 10^3/uL
Arm/Group | Autologous Blood Transfusion | Allogenic Blood Transfusion
Number analyzed (Participants) | 20 | 25
10^3/uL | 7.2 (1.7) | 5.7 (1.5)

37. Secondary Outcome: Lymphocytes
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: percentage of white blood cells
Arm/Group | Autologous Blood Transfusion | Allogenic Blood Transfusion
Number analyzed (Participants) | 20 | 25
percentage of white blood cells | 38.3 (13) | 47.3 (14)

38. Secondary Outcome: Lymphocytes
Time Frame: Day 1 postop
Measure: Mean (Standard Deviation); unit: percentage of white blood cells
Arm/Group | Autologous Blood Transfusion | Allogenic Blood Transfusion
Number analyzed (Participants) | 20 | 25
percentage of white blood cells | 22.7 (11) | 24.3 (11)

39. Secondary Outcome: Lymphocytes
Time Frame: Day 5 postop
Measure: Mean (Standard Deviation); unit: percentage of white blood cells
Arm/Group | Autologous Blood Transfusion | Allogenic Blood Transfusion
Number analyzed (Participants) | 20 | 25
percentage of white blood cells | 33.3 (12) | 36.1 (11)

40. Secondary Outcome: Lymphocytes
Time Frame: Day 8 postop
Measure: Mean (Standard Deviation); unit: percentage of white blood cells
Arm/Group | Autologous Blood Transfusion | Allogenic Blood Transfusion
Number analyzed (Participants) | 20 | 25
percentage of white blood cells | 33.6 (7) | 42.5 (11)

ADVERSE EVENTS:
Arm/Group | Autologous Blood Transfusion | Allogenic Blood Transfusion
Serious Adverse Events (participants affected / at risk) | 0/20 | 2/25
Other Adverse Events (participants affected / at risk) | 10/20 | 8/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Autologous Blood Transfusion (N=20) | Allogenic Blood Transfusion (N=25)
Haemoarthrosis of the operated knee (Musculoskeletal and connective tissue disorders) | 0 (0) | 1/1 (1)
Crural phlebothrombosis of the operated limb (Vascular disorders) | 0 (0) | 1/1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Autologous Blood Transfusion (N=20) | Allogenic Blood Transfusion (N=25)
Fever (General disorders) | 4 (4) | 5 (5)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 2 (2) | 1 (1)
Constipation (Metabolism and nutrition disorders) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days